CLINICAL TRIAL: NCT05815732
Title: HEBE - Healthy Aging Versus Inflamm-aging: the Role of Physical Exercise in Modulating the Biomarkers of Age-associated and Environmentally Determined Chronic Diseases. Research Line 1. Proof of Concept
Brief Title: HEBE Project - Healthy Aging Versus Inflamm-aging: the Role of Physical Exercise in Modulating the Biomarkers of Age-associated and Environmentally Determined Chronic Diseases
Acronym: HEBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Milan (Other)
Collaborators: Istituto Auxologico Italiano (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Elia Mario Biganzoli, Full Professor of Medical Statistics, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HEBE
Record Dates: First submitted 2023-03-01; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Aging
Keywords: chronic inflammation; physical exercise; lifestyle; prevention
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be assessed before and after the intervention with physical exercise and personalized lifestyle advice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercise prescription (Experimental): Prescription of a personalized exercise program, which will define modalities, intensity, duration, frequency and progression of the exercise. For each subject, at baseline and after 6 months, biological samples will be collected (blood, urine, saliva and nasal swab)
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Personalized exercise program, with defined modalities, intensity, duration, frequency and progression of the exercise.

SUMMARY:
The main objective of this clinical trial is to test the effects of the personalized intervention based on physical exercise, on clinical variables and circulating markers, in a population of employees of the University of Milan (UMilan).

The HEBE study will include two phases:

PHASE 1:

All UMilan employees will be asked to voluntarily complete an anonymous online questionnaire, in order to gather information about their lifestyle (physical activity, diet, cigarette smoking, etc) (zero time: T0); at the end of the compilation, indications on how to improve the lifestyle will be provided. These indications will also be present and available for consultation in a special section of the site on the "HEBE" site, with UMilan domain (www.hebe.unimi.it).

After 6 months, all UMilan employees will receive a second invitation to voluntarily complete the same questionnaire, in order to evaluate any changes, in terms of lifestyle improvement (time one: T1).

PHASE 2:

100 eligible subjects who have expressed their availability in the initial questionnaire, will be identified to undergo a lifestyle improvement protocol based mainly on the prescription of a personalized exercise program, which will define modalities, intensity, duration, frequency and progression of the exercise. For each subject, at T0 and T1 (after 6 months), biological samples will be collected (blood, urine, saliva and nasal swab), which will be used to: i) set up a biobank shared by the members of the HEBE consortium; ii) identify biomarkers able to monitor the effect of physical exercise on the characteristics of the frailty under examination. Furthermore, both at T0 and T1 questionnaires will be completed and carried out clinical evaluations (anamnesis, physical examination, tests for the study of the autonomic nervous system, bio-impedance test, evaluation/estimate of maximal oxygen consumption, ECG).

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) are the cause of premature aging and death of 41 million people each year, accounting for 71% of all deaths globally. NCDs are closely linked to rapid urbanization and globalization. In this context, unsustainable lifestyles, characterized by a lack of physical activity, trigger the progression of NCDs. To date, it is estimated that around 41% of Europeans (and as many as 60% of Italians) do not engage in any type of physical activity (even light) during the week and this increases the risk of chronic diseases: 86% of deaths are attributable to cardiovascular disease, cancer, chronic respiratory disease and type 2 diabetes, a disease from which approximately 52 million people suffer in Europe (8.4% of men and 7.8% of women among 20 and 79 years of age).

Over the years, the progressive increase in the number of senescent cells can lead to tissue/organ dysfunction. In an attempt to respond to this process, senescent cells undergo metabolic modifications leading to increased secretion of soluble factors (e.g. cytokines, chemokines, growth factors, metalloproteases), which thus modulate their microenvironment through the removal of damaged cells by the recruitment of phagocytes and stimulating cell differentiation and proliferation for tissue renewal. The secretion of pro-inflammatory molecules and the activation of immune cells contributes to the generation of a low-grade chronic pro-inflammatory state known as "inflammaging", which is at the root of most age-related diseases. Furthermore, upregulation of mitogenic and pro-angiogenic pathways dangerously increases the risk of oncogenic transformation. The modulation of the complex of alterations that make up inflammaging could therefore be the key to guaranteeing healthy aging and reducing the risk of developing early NCD. A very promising approach to controlling inflammaging involves focusing on reducing the risk factors associated with these diseases by proposing alternative development models.

The main challenge of the HEBE project as a whole therefore consists in addressing three fundamental questions:

1. What primary prevention approaches can we develop, considering all phases of the individual's life, to ensure an improvement in the quality of life and health status of the population, with a positive impact on the socio-economic system of the area?
2. What intervention protocols based on physical exercise, combined with diet and any pharmacological/pharmaceutical approach, can we propose to frail subjects, in order to intervene on "inflammaging", to increase life expectancy and healthy ageing?
3. Which inflammaging markers (biomarkers and other clinical indicators) can we measure and integrate to define the risk of developing NCD, especially in frail subjects, to guide integrated personalized preventive interventions (precision/personalized healthcare)?

General objectives of the trial

The main objective of this study is the evaluation of the effects of the personalized intervention based on physical exercise, on clinical parameters and circulating markers, in a population of employees of the University of Milan (UMilan).

In Research Line 1- a pilot study will be conducted involving UMilan employees which will include two phases:

PHASE 1:

All UMilan employees will be asked to voluntarily complete an anonymous online questionnaire, in order to gather information about their lifestyle (physical activity, diet, cigarette smoking, etc.) (zero time: T0); at the end of the compilation, indications on how to improve the lifestyle will be provided. These indications will also be present and available for consultation in a special section of the site on the "HEBE" site, with UMilan domain (www.hebe.unimi.it), in a special section.

After 6 months, all UMilan employees will receive a second invitation to voluntarily complete the same questionnaire, in order to evaluate any changes, in terms of lifestyle improvement (time one: T1).

PHASE 2:

100 eligible subjects who have expressed their availability in the initial questionnaire, will be identified to undergo a lifestyle improvement protocol based mainly on the prescription of a personalized exercise program, which will define modalities, intensity, duration, frequency, and progression of the exercise. For each subject, at T0 and T1 (after 6 months), biological samples will be collected (blood, urine, saliva and nasal swab), which will be used to: i) set up a biobank shared by the members of the HEBE consortium; ii) identify biomarkers able to monitor the effect of physical exercise on the characteristics of the frailty under examination. Furthermore, both at T0 and T1 questionnaires will be completed and carried out clinical evaluations (anamnesis, physical examination, tests for the study of the autonomic nervous system, bio-impedance test, evaluation/estimate of maximal oxygen consumption, ECG) useful for: i) verifying the clinical conditions of the subject; ii) obtain useful parameters for the customized definition of the intervention program; iii) verify the effectiveness of the intervention at T1; iv) assess the association between clinical indicators and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Being an employee of UMilan of both sexes and of any age (18-70 years);
* For the 100 chosen subjects identified for Phase 2: declare that they do not carry out physical activities at a competitive level and that you are committed about improving your own lifestyle.

Exclusion Criteria:

* Previous myocardial infarction
* Autoimmune diseases
* Neurodegenerative pathologies
* Psychiatric pathologies
* Cardiac arrhythmias
* Chronic obstructive pulmonary disease
* osteo-muscular problems that prevent the execution of physical activity;
* oncological pathologies in the last 3 years that have required chemotherapy or immunotherapy;
* pregnancy/nursing/intention to become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in maximal oxygen consumption (VO2 max) | Change from baseline VO2 max at six months
  The maximum or optimum rate at which the heart, lungs, and muscles can effectively use oxygen during exercise, used as a way of measuring a person's individual aerobic capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Elia M Biganzoli, PhD, Study Director — University of Milan; Daniela Lucini, PhD, Principal Investigator — University of Milan; Valentina Bollati, PhD, Principal Investigator — University of Milan; Francesca Bianchi, PhD, Principal Investigator — University of Milan; Chiara Mandò, PhD, Principal Investigator — University of Milan; Mario Clerici, PhD, Study Chair — University of Milan
Locations (1):
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The plan is going to be agreed with all the 140 participants Researchers of UMilan of the HEBE project with a Consortium Agreement

REFERENCES:
- [Derived] Bianchi F, Biganzoli EM, Bollati V, Clerici M, Lucini D, Mando C, Rota F; HEBE Consortium. HEBE project: Healthy aging versus inflamm-aging: The role of physical exercise in modulating the biomarkers of age-associated and environmentally determined chronic diseases, study protocol. PLoS One. 2024 Apr 30;19(4):e0300011. doi: 10.1371/journal.pone.0300011. eCollection 2024. PMID 38687742
- See also: HEBE project website — https://hebe.unimi.it/